CLINICAL TRIAL: NCT02979951
Title: An International, Multicentre, Non-comparative, Non-interventional, Prospective Clinical Registry to Evaluate the Clinical Outcome and Safety of the Treatment of Severely Infected Patients with Fosfomycin I.v.
Brief Title: Fosfomycin I.v. for Treatment of Severely Infected Patients
Acronym: FORTRESS
Status: Recruiting | Type: Observational
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: INPADS GmbH (Unknown); Dr. Oestreich + Partner GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: FORTRESS
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Infections; Bone Diseases, Infectious; Osteomyelitis; Central Nervous System Bacterial Infections; Meningitis, Bacterial; Encephalitis; Brain Abscess; Urinary Tract Infections; Respiratory Tract Infections; Pneumonia, Bacterial; Skin Diseases, Bacterial; Soft Tissue Infections; Intraabdominal Infections; Sepsis; Bacteremia; Endocarditis, Bacterial
Keywords: Observational Study; Non-Interventional Study; Registries; Prospective; Monitored; Multicentric; International; Fosfomycin; Infectofos; Fomicyt; Bacterial Infections; Gram-Negative Bacterial Infections; Gram-Positive Bacterial Infections; Bone Diseases, Infectious; Osteomyelitis; Central Nervous System Bacterial Infections; Meningitis, Bacterial; Encephalitis; Brain Abscess; Urinary Tract Infections; Respiratory Tract Infections; Pneumonia, Bacterial; Skin Diseases, Bacterial; Soft Tissue Infections; Intraabdominal Infections; Sepsis; Bacteremia; Endocarditis, Bacterial; Treatment Outcome; Clinical Efficacy; Microbiological Efficacy; Safety
MeSH Terms: conditions — Bacterial Infections; Bone Diseases, Infectious; Osteomyelitis; Central Nervous System Bacterial Infections; Meningitis, Bacterial; Encephalitis; Brain Abscess; Urinary Tract Infections; Respiratory Tract Infections; Pneumonia, Bacterial; Skin Diseases, Bacterial; Soft Tissue Infections; Intraabdominal Infections; Sepsis; Bacteremia; Endocarditis, Bacterial; Gram-Negative Bacterial Infections; Gram-Positive Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this European, multicentric, prospective, non-interventional study is to document and evaluate the efficacy and safety of the treatment of severely infected patients with intravenously administered fosfomycin, including patients with osteomyelitis, complicated urinary tract infection, nosocomial lower respiratory tract infection, bacterial meningitis/central nervous system infection, bacteraemia/sepsis, skin and soft tissue infection, endocarditis or other infections, each as far as covered by the respective nationally relevant SmPC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years
* Treatment with fosfomycin according to the (national) Summary of Product Characteristics (SmPC) of fosfomycin i.v.
* Patients with osteomyelitis, complicated urinary tract infection, nosocomial lower respiratory tract infection, bacterial meningitis/central nervous system infection, bacteraemia/sepsis, skin and soft tissue infection, endocarditis or other infection, each as far as covered by the respective nationally relevant SmPC
* Written informed consent of the participant (or person in charge in case of patients incapable of giving consent)

Exclusion Criteria:

* Previous documentation of the patient in the present study
* Patients participating in an interventional clinical trial
* Patients with known hypersensitivity to fosfomycin or any of the excipients
* Terminally ill patients
* Patients with "do not resuscitate order"
* Palliative treatment approach
* Failure of > 3 of the following organ systems: respiratory system, nervous system, cardiovascular system, liver, coagulation, kidney
* Manifest Human Immunodeficiency Virus (HIV) disease (Acquired Immunodeficiency Syndrome, AIDS)
* Fosfomycin treatment as 4th line treatment or at later stage
* Patients with involvement of fungi or mycobacteria in the targeted infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of the participating study sites (clinics specialised and experienced in the management and treatment of patients suffering from (a part of) the included diseases as mentioned in the respective inclusion criterion), who fulfill all inclusion criteria and do not fulfill any of the exclusion criteria, are eligible for participation in the FORTRESS study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-12; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with clinical success as defined as clinical cure or clinical improvement | Analysed at EOT ("End of fosfomycin treatment", up to 6 months after start of fosfomycin treatment)
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "End of fosfomycin treatment" (EOT) is reached at the day of the last fosfomycin application in the course of the treatment schedule for the targeted infection (i.e., in case of a multiple stage treatment schedule, the end of the last fosfomycin treatment phase).

SECONDARY OUTCOMES:
Microbiological cure | Analysed at "initial response" (not later than 7 days after start of fosfomycin treatment)
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "initial response" is defined to be after start of fosfomycin treatment and not later than 7 days after start of fosfomycin treatment.
Microbiological cure | Analysed at EOT ("End of fosfomycin treatment", up to 6 months after start of fosfomycin treatment)
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "End of fosfomycin treatment" (EOT) is reached at the day of the last fosfomycin application in the course of the treatment schedule for the targeted infection (i.e., in case of a multiple stage treatment schedule, the end of the last fosfomycin treatment phase).
Microbiological cure | Analysed at TOC ("Test of cure", up to 6 months after start of fosfomycin treatment)
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "TOC" is defined to be not earlier than EOT and not later than end of hospital stay of the patient.
Microbiological cure | Analysed at follow-up (within one year after start of fosfomycin treatment) (only for indication "osteomyelitis")
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Defined to be after end of hospital stay + within 1 year after start of fosfomycin treatment. Either the latest visit after "End of hospital stay" within 1 year after start of fosfomycin treatment or, if applicable, the visit in this time frame assessing a clinical failure/relapse.
Clinical success as defined as clinical cure or clinical improvement | Analysed at "initial response" (not later than 7 days after start of fosfomycin treatment)
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "initial response" is defined to be after start of fosfomycin treatment and not later than 7 days after start of fosfomycin treatment.
Clinical success as defined as clinical cure or clinical improvement | Analysed at TOC ("Test of cure", up to 6 months after start of fosfomycin treatment)
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "TOC" is defined to be not earlier than EOT and not later than end of hospital stay of the patient.
Clinical success as defined as clinical cure or clinical improvement | Analysed at follow-up (within one year after start of fosfomycin treatment) (only for indication "osteomyelitis")
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Defined to be after end of hospital stay + within 1 year after start of fosfomycin treatment. Either the latest visit after "End of hospital stay" within 1 year after start of fosfomycin treatment or, if applicable, the visit in this time frame assessing a clinical failure/relapse.
Clinical cure | Analysed at EOT ("End of fosfomycin treatment", up to 6 months after start of fosfomycin treatment)
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "End of fosfomycin treatment" (EOT) is reached at the day of the last fosfomycin application in the course of the treatment schedule for the targeted infection (i.e., in case of a multiple stage treatment schedule, the end of the last fosfomycin treatment phase).
Clinical cure | Analysed at TOC ("Test of cure", up to 6 months after start of fosfomycin treatment)
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "TOC" is defined to be not earlier than EOT and not later than end of hospital stay of the patient.
Clinical cure | Analysed at follow-up (within one year after start of fosfomycin treatment) (only for indication "osteomyelitis")
  Definition of clinical cure (both criteria must be fulfilled):
  * Resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Defined to be after end of hospital stay + within 1 year after start of fosfomycin treatment. Either the latest visit after "End of hospital stay" within 1 year after start of fosfomycin treatment or, if applicable, the visit in this time frame assessing a clinical failure/relapse.
Clinical improvement | Analysed at "initial response" (not later than 7 days after start of fosfomycin treatment)
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "initial response" is defined to be after start of fosfomycin treatment and not later than 7 days after start of fosfomycin treatment.
Clinical improvement | Analysed at EOT ("End of fosfomycin treatment", up to 6 months after start of fosfomycin treatment)
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "End of fosfomycin treatment" (EOT) is reached at the day of the last fosfomycin application in the course of the treatment schedule for the targeted infection (i.e., in case of a multiple stage treatment schedule, the end of the last fosfomycin treatment phase).
Clinical improvement | Analysed at TOC ("Test of cure", up to 6 months after start of fosfomycin treatment)
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Time point "TOC" is defined to be not earlier than EOT and not later than end of hospital stay of the patient.
Clinical improvement | Analysed at follow-up (within one year after start of fosfomycin treatment) (only for indication "osteomyelitis")
  Definition of clinical improvement (both criteria must be fulfilled):
  * Partial resolution of signs and symptoms and
  * microbiological cure or no additional antibiotic therapy for the targeted infection necessary.
  Definition of microbiological cure:
  * Elimination of the relevant pathogen(s) at the relevant site(s) of infection (at least one negative culture) or
  * in case "no sample available/indicated due to sufficient clinical response", pathogen elimination is considered.
  Time Frame:
  Defined to be after end of hospital stay + within 1 year after start of fosfomycin treatment. Either the latest visit after "End of hospital stay" within 1 year after start of fosfomycin treatment or, if applicable, the visit in this time frame assessing a clinical failure/relapse.
Sodium serum levels | On every day from start of fosfomycin treatment until end of hospital stay (up to 6 months after start of fosfomycin treatment)
Potassium serum levels | On every day from start of fosfomycin treatment until end of hospital stay (up to 6 months after start of fosfomycin treatment)
Adverse events | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)
Non-serious adverse events | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)
Serious adverse events | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)
Cases of death | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)
Adverse drug reactions (ADRs) | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)
Serious adverse drug reactions (SADRs) | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)
Dropouts due to treatment failure or due to adverse events | On every day from start of fosfomycin treatment until end of follow-up (up to one year after start of fosfomycin treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus-Friedrich Bodmann, Dr., Study Director — Klinik Nordoberpfalz AG, Klinikum Weiden
Locations (50):
- Austria (4):
  - Landeskrankenhaus Hall - Tirol Kliniken, Hall in Tirol
  - A.ö. Bezirkskrankenhaus, Reutte
  - AKH Wien, Universitätsklinik für Innere Medizin 1, Vienna
  - Klinikum Wels-Grieskirchen, Institut für Hygiene und Mikrobiologie, Wels
- Germany (14):
  - Universitätsmedizin Charité, Berlin
  - Vivantes Kliniken Neukölln, Berlin
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Universitäts Düsseldorf; Klinik für Anästhesiologie, Düsseldorf
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universität Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena; Zentrum für Infektionsmedizin, Jena
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinik Schleswig-Holstein, Lübeck
  - LMU München, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Oldenburg, Oldenburg in Holstein
  - Universitätsklinik Regensburg; Klinik für Anästhesiologie, Regensburg
  - Kliniken Nordoberpfalz, Weiden
- Greece (11):
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Kifissia, Athens
  - General Hospital of Athens "Evangelismos", Athens
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - University General Hospital "ATTIKON", Athens
  - General Hospital of Attica "KAT", Kifissia
  - General Hospital of Lamia, Lamia
  - RIO Univ. Hospital, Dept of Pathology, Division of Infectious Diseases, Pátrai
  - "AHEPA" University General Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G. GENIMMATAS", Thessaloniki
  - General Hospital of Thessaloniki "Hippokration", Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- Italy (12):
  - Clinical Malattie Infettive, Bari
  - Azienda Ospedaliera S.Croce e Carle, Cuneo
  - Ospedal Policlinico San Martino, Genova
  - Ospedale L. Sacco, Milan
  - Istituto Mediterraneo per i Trapianti Ismett IRCCS, Palermo
  - Policlinico Paolo Giaccone, Palermo
  - Policlinico Umberto I, Malattie Infettive, Rome
  - Lazzaro Spallanzani, Rome
  - Polocinico Tor Vergata, Rome
  - AOU Città della Salute e Scienza-Presidio Molinette, Torino
  - Ospedale S.M.della Misericordia, Udine
  - ASST-Sette Lagh Viale Borre, Varese
- United Kingdom (9):
  - Royal Bolton Hospital, Bolton
  - Hull & East Yorkshire Hospitals NHS Trust, Cottingham
  - Ninewells Hospital, Dundee
  - Queen Elisabeth University Hospital, Glasgow
  - University of Glasgow/Royal Infirmary, Glasgow
  - University Hospital Crosshouse, Kilmarnock
  - Chelsea & Westminster Hospial, London
  - Queen Elisabeth Hospital, London
  - Univresity College Londen (UCL) Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bodmann KF, Hagel S, Oliva A, Kluge S, Mularoni A, Galfo V, Falcone M, Pletz MW, Lindau S, Kading N, Kielstein JT, Zoller M, Tascini C, Kintrup S, Schadler D, Spies C, De Rosa FG, Radnoti S, Bandera A, Luzzati R, Allen S, Sarmati L, Cascio A, Kapravelos N, Subudhi CPK, Dimopoulos G, Vossen MG, Bal AM, Venditti M, Mastroianni CM, Borrmann T, Mayer C. Real-World Use, Effectiveness, and Safety of Intravenous Fosfomycin: The FORTRESS Study. Infect Dis Ther. 2025 Apr;14(4):765-791. doi: 10.1007/s40121-025-01125-2. Epub 2025 Mar 19. PMID 40106180